CLINICAL TRIAL: NCT02353117
Title: Preventing Congenital Syphilis
Acronym: PCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Public Health and Tropical Medicine (Other)
Collaborators: Instituto de Efectividad Clinica y Sanitaria (IECS) (Unknown); Kinshasa School of Public Health (Other); University of Zambia (Other)
Responsible Party: Principal Investigator, Dr. Pierre Buekens, W.H. Watkins Professor and Dean, Tulane University
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPP1116131
Record Dates: First submitted 2015-01-21; First posted 2015-02-02 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Congenital Syphilis
MeSH Terms: conditions — Syphilis, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Behavioral intervention. The intervention will be multifaceted, tailored by formative research, and include: 1) opinion leaders, reminders, monitoring, and feedback; 2) point-of-care rapid tests and immediate treatment if the rapid test is positive; and 3) locally packaged treatment kits (benzathine penicillin 2.4 MIU, syringe and needle, instructions, and information on side-effects).
  Interventions: Behavioral: Congenital Syphilis Intervention Group
- Control (No Intervention): Prenatal care providers at control clinics will be invited to participate in a training workshop. They will be given refresher concepts on the prenatal care package and maternal and congenital syphilis and will be trained in syphilis case detection and management, using their standard and available screening methods. They will also be trained on how to document the screening and treatment process, using the same system as the intervention clinics. No other activities are planned in the control group; providers will be encouraged to disseminate and implement any strategy they consider useful to improve screening and treatment. Study personnel will ensure the availability of screening tests already in-use, as well as ensure the availability of benzathine penicillin at all control prenatal clinics.

INTERVENTIONS:
Behavioral: Congenital Syphilis Intervention Group
  Arms: Intervention

SUMMARY:
Nearly 1.5 million pregnant women are infected with syphilis each year, and it is estimated that half of them will have adverse birth outcomes. Congenital syphilis remains a major public health issue, despite the fact that maternal syphilis is easy to detect and treat. Multiple barriers impair the elimination of congenital syphilis. Syphilis is often stigmatized and of low priority, and even women attending prenatal care early are potentially facing multiple clinical barriers. The study objective is to use implementation research methods to evaluate a multifaceted intervention to increase the use of evidence-based clinical procedures to prevent congenital syphilis. The investigators will perform a facility-based, two-arm parallel cluster randomized implementation trial in the Democratic Republic of the Congo and Zambia. The intervention will be multifaceted, tailored by formative research, and include: opinion leaders, reminders, monitoring, and feedback; point-of-care rapid tests; and treatment kits to be used immediately if the rapid test is positive. Improving syphilis screening and treatment will be promoted as a key step toward improving the quality of all components of prenatal care.

DETAILED DESCRIPTION:
Scope:

The investigators will use implementation research methods to evaluate a multifaceted intervention to increase the use of evidence-based clinical procedures to prevent congenital syphilis. Improving syphilis screening and treatment will be promoted as a key step toward improving the quality of all components of prenatal care.

The objective is to increase the frequency of pregnant women attending prenatal care screened for syphilis and treated if infected (primary outcomes). The investigators will also measure the impact of the intervention on other components of prenatal care (screening for anemia, HIV, proteinuria) (secondary outcomes).

Approach:

Design: Facility-based, two-arm parallel cluster randomized implementation trial. Clusters correspond to geographic areas with several prenatal clinics. After a six-month period of baseline data collection, clusters will be randomized to either an intervention group or a control group. For 18 months, the prenatal clinics in the intervention clusters will conduct the multifaceted intervention. The prenatal clinics in the control clusters will continue their usual activities. Data collected during the intervention period will be compared to baseline data.

Sample Size: The investigators are assuming that 300 women will initiate prenatal care per cluster each year. A sample size of 20 clusters (10 per arm) with three women seropositive for syphilis per cluster will achieve more than 80% power to detect an increase in treated women from 50% to 85%, with a significance level of the test of 0.05, and an intracluster correlation coefficient of 0.01. This will give more than 90% power to detect an increase in the number of women with a complete screening from 50% to 75%. Calculations are based on the conservative assumption that 50% of women are screened and 50% are treated at baseline; lower screening and treatment rates at baseline would increase the power of the proposed study.

Settings: DRC (10 clusters), Zambia (10 clusters), and Argentina (Data Center).

* In the DRC, the study will be performed in the Maluku and Nsele health areas, which are located within the capital city-province of Kinshasa.
* In Zambia, the study will be performed in the health areas of Kafue and Chongwe, which are located within the capital province of Lusaka.
* The Data Center will be located in Buenos Aires, Argentina.

Intervention: The intervention will be multifaceted, tailored by formative research, and include:

1. Opinion leaders, reminders, monitoring, and feedback;
2. Point-of-care rapid tests and immediate treatment if the rapid test is positive;
3. Locally packaged treatment kits (benzathine penicillin 2.4 MIU, syringe and needle, instructions, and information on side-effects).

Even though screening and treatment should occur as early as possible during pregnancy, benefit is expected at any stage of pregnancy. No woman will be excluded based on gestational age.

Opinion leaders in the intervention prenatal clinics will be identified by their peers and invited to work as "facilitators." Training will include: the content of the prenatal care package recommended by WHO and the need to improve the quality of all components of prenatal care; the importance of maternal and congenital syphilis and case management based on WHO recommendations; screening with point-of-care rapid tests and same-day treatment for those found positive; managing allergies to penicillin; how to ensure that all pregnant women are screened; and how to conduct one-on-one detailing visits with prenatal clinic providers to discuss their views regarding the implementation of the screening and treatment program.

After completing the training, the facilitators will return to their prenatal clinics to implement the program, which will include training other prenatal care providers and conducting personal visits with each of them to discuss their perspectives and potential barriers. The facilitators will be responsible for placing the treatment kits in convenient sites to ensure ease of use in infected women and for developing simple reminders to be placed in consultation offices and patient waiting areas. The facilitator teams will also produce periodical reports on the rates of syphilis screening and treatment and will distribute these reports to all prenatal care providers. Cluster coordinators will meet periodically with each team to assess the completion of activities and to address unexpected problems. The intervention will be refined, taking into account the information obtained during the formative research phase. Thus, the components described above may be modified after the formative research stage.

Activities at Control Clinics: As a standard training procedure, prenatal care providers at control clinics will be invited to participate in a half-day training workshop. They will be given refresher concepts on the prenatal care package and maternal and congenital syphilis and will be trained in syphilis case detection and management, using their standard and available screening methods. Additionally, they will be trained on how to document the screening and treatment process, using the same system as the intervention clinics. No other activities are planned in the control group, but prenatal care providers will be encouraged to disseminate and implement any strategy they consider useful to improve the screening and treatment process. Study personnel will ensure the availability of screening tests already in-use, as well as ensure the availability of benzathine penicillin at all control prenatal clinics.

ELIGIBILITY:
Inclusion Criteria: Pregnant women who present for prenatal care at a participating prenatal care clinic for the first time who consent to participate in the study.

Exclusion Criteria: Pregnant women who do not agree to participate in the study.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60386 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
The frequency of pregnant women attending prenatal care screened for syphilis and treated if infected | 18 months

SECONDARY OUTCOMES:
The number of women who receive screening for other components of prenatal care (anemia, HIV, proteinuria). | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Buekens, MD, PhD, Principal Investigator — Tulane SPHTM
Locations (4):
- Tulane School of Public Health and Tropical Medicine, New Orleans, Louisiana, United States
- Institute for Clinical Effectiveness and Health Policy, Buenos Aires, Argentina
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo
- University Teaching Hospital, University of Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Althabe F, Chomba E, Tshefu AK, Banda E, Belizan M, Bergel E, Berrueta M, Bertrand J, Bose C, Cafferata ML, Carlo WA, Ciganda A, Donnay F, Garcia Elorrio E, Gibbons L, Klein K, Liljestrand J, Lusamba PD, Mavila AK, Mazzoni A, Nkamba DM, Mwanakalanga FH, Mwapule Tembo A, Mwenechanya M, Pyne-Mercier L, Spira C, Wetshikoy JD, Xiong X, Buekens P. A multifaceted intervention to improve syphilis screening and treatment in pregnant women in Kinshasa, Democratic Republic of the Congo and in Lusaka, Zambia: a cluster randomised controlled trial. Lancet Glob Health. 2019 May;7(5):e655-e663. doi: 10.1016/S2214-109X(19)30075-0. Epub 2019 Mar 22. PMID 30910531